CLINICAL TRIAL: NCT00967278
Title: Hemodynamic Changes in Off-pump Coronary Artery Bypass Grafting
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Maria José Carvalho Carmona, University of Sao Paulo
Other Study IDs: FAPESP 03/07092-6
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Coronary Artery Disease
Keywords: OPCAB; pulmonary artery catheter; esophageal doppler; hemodynamics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Off-Pump: Patients with coronary artery disease undergoing elective off-pump CABG

SUMMARY:
The purpose of this study is to study the positioning and stabilization of different cardiac walls performed during off-pump coronary artery bypass grafting (CABG) may have dissimilar impact on hemodynamics.

The objective is to evaluate hemodynamics during distal coronary anastomoses in different cardiac walls.

DETAILED DESCRIPTION:
* Twenty patients undergoing off-pump CABG monitored with pulmonary artery catheter and esophageal doppler will be enrolled.
* Patients with a left ventricular ejection fraction <50%, age >80 yr, creatinine >1.4 mg/dl, reoperation, valvular heart disease or chronic obstructive pulmonary disease were excluded
* Data will be collected after volemic and hemodynamic adjustments, after heart positioning and establishment of a suction stabilizer and before its removal in anterior, lateral or posterior wall artery anastomosis.
* Data was compared by means of two-way repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Normal left ventricular function
* Minimal to moderate surgical risk according to criteria proposed by Higgins et al. (JAMA. 1992 May 6;267(17):2344-8)

Exclusion Criteria:

* Patients with a left ventricular ejection fraction <50%,
* Age >80 yr
* Creatinine >1.4 mg/dl
* Reoperation
* Valvular heart disease
* Chronic obstructive pulmonary disease
* High surgical risk according to criteria proposed by Higgins et al. (JAMA. 1992 May 6;267(17):2344-8)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with coronary artery disease indicated to elective surgical treatment
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil